CLINICAL TRIAL: NCT02921698
Title: Safety and Efficacy Analysis of FRED® Embolic Device in Aneurysm Treatment
Acronym: SAFE
Status: Completed | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SAFE
Record Dates: First submitted 2016-09-27; First posted 2016-10-03 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2017-08

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- FRED®
  Interventions: Device: FRED®

INTERVENTIONS:
Device: FRED® — Flow Re-Direction Endoluminal Device

SUMMARY:
A prospective, multicenter, observational evaluation of the safety and efficacy of the FRED® device in the treatment of intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is aged ≥18 years
2. Patient has an unruptured or recanalized intracranial aneurysm :

   * for which an endovascular treatment has been determined appropriate
   * that can not be treated by standard techniques (coiling with or without remodeling)
   * and for which the FRED® Flow Diverter has been determined an appropriate treatment
3. Patient or patient's legally authorized representative has been informed about the confidentiality of the study and agrees to the collection of his/her personal data
4. Patient presents with an mRS score between 0 and 2
5. Patients who have already been treated with a stent or a flow diverter for another aneurysm may be included if:

   * the previous treatment was more than three months prior to enrollment in this study
   * the aneurysm to be treated for this study is a new aneurysm located on a different parent vessel unless the stent already in place is implanted on the proximal carotid artery.

Exclusion Criteria:

1. Patient has a known allergy to antiplatelet therapy, heparin and/or contrast medium
2. Patient has contraindication to antiplatelet therapy and/or heparin
3. Patient is pregnant and/or breastfeeding
4. Patient may not benefit from imaging and clinical monitoring
5. Patient has a medical or surgical co-morbidities limiting his/her life expectancy to less than 1 year
6. Patient will be treated with a flow diverter other than FRED®
7. Patient had an intracranial hemorrhage within the 30 days preceding treatment
8. Patient has an aneurysm(s) with one or more of the following characteristics:

   * associated with an arteriovenous malformation
   * dissecting or ""blister-like""
   * multiple (unless only one aneurysm requires treatment)
   * located in the posterior circulation
   * treated with a stent or a flow diverter on the same parent vessel (excluding proximal carotid artery) or in the 3 months prior to inclusion
9. Patient has stenosis of the aneurysm parent artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged a minimum of 18 years with an unruptured or recanalized intracranial aneurysm in whom endovascular treatment has been determined the appropriate treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2017-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Aneurysm occlusion without ˃ 50% parent artery stenosis | 6 months
Morbidity rate | 6 months
Mortality rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pierot, Prof., Principal Investigator — CHU Reims; Reims, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pierot L, Spelle L, Berge J, Januel AC, Herbreteau D, Aggour M, Piotin M, Biondi A, Barreau X, Mounayer C, Papagiannaki C, Lejeune JP, Gauvrit JY, Derelle AL, Chabert E, Costalat V. SAFE study (Safety and efficacy Analysis of FRED Embolic device in aneurysm treatment): 1-year clinical and anatomical results. J Neurointerv Surg. 2019 Feb;11(2):184-189. doi: 10.1136/neurintsurg-2018-014261. Epub 2018 Oct 8. PMID 30297539
- [Derived] Pierot L, Spelle L, Berge J, Januel AC, Herbreteau D, Aggour M, Piotin M, Biondi A, Barreau X, Mounayer C, Papagiannaki C, Lejeune JP, Gauvrit JY, Costalat V. Feasibility, complications, morbidity, and mortality results at 6 months for aneurysm treatment with the Flow Re-Direction Endoluminal Device: report of SAFE study. J Neurointerv Surg. 2018 Aug;10(8):765-770. doi: 10.1136/neurintsurg-2017-013559. Epub 2018 Jan 19. PMID 29352057